CLINICAL TRIAL: NCT07202637
Title: Evaluation of the Variation of the Sub-pulmonary Velocity-time Integral to Predict Fluid Responsiveness Prospective Observational Study
Brief Title: Evaluation of the Variation of the Sub-pulmonary Velocity-time Integral to Predict Fluid Responsiveness
Status: Recruiting | Type: Observational
Sponsor: Hospital Nord (Other)
Responsible Party: Principal Investigator, Gary DUCLOS, MD, MSc, Aix Marseille Université
Other Study IDs: ITV-VD; 2023-A02636-39 (Other: Comité de protection des personnes - Ouest I)
Record Dates: First submitted 2025-09-12; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fluid Resuscitation; Fluid Responsiveness Predictability
Keywords: fluid responsiveness; echocardiography; Passive Leg Raising; Mini Fluid Challenge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suspected of hypovolemia: Patients with suspected hypovolemia who need to be evaluated for fluid responsiveness
  Interventions: Drug: Fluid bolus administration

INTERVENTIONS:
Drug: Fluid bolus administration — Fluid infusion of 500 mL of a crystalloïd solution is performed for patients with signs of hypovolemia

SUMMARY:
Fluid administration is the first-line treatment in hypovolemic states in critically ill patients. Prediction of fluid responsiveness is possible with echocardiography by assessing the variation of the sub-aortic velocity-time integral (AoVTI) during a passive leg raising test (PLR) or Mini-fluid challenge. However, VTI-Ao measurement is not feasible in all patients due to poor echogenicity. Validation of new fluid-responsiveness indices may facilitate the evaluation in this patient population. Among the available indices, variation of the sub-pulmonary VTI is a potential criterion.

ELIGIBILITY:
Inclusion Criteria:

* Patient with measurable sub-pulmonary VTI in at least one of the two windows: parasternal short-axis or subcostal.
* Patient with measurable sub-aortic VTI in apical 4-chamber view before and after PLR maneuver.
* Patient with suspected hypovolemia or whose hemodynamic status justifies vasopressor infusion.

Exclusion Criteria:

* Severe left ventricular dysfunction defined by left ventricular ejection fraction (LVEF) < 30%.
* Severe right ventricular dysfunction defined by TAPSE < 12 mm.
* Cardiac arrhythmia or atrial fibrillation.
* Abdominal compartment syndrome.
* Amputation of one or both lower limbs.
* Intracranial hypertension.
* Pregnant women (ruled out by systematic pregnancy test at ICU admission).
* Minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In patients with suspected hypovolemia, a cardiac ultrasound is performed as part of routine care. A patient is eligible if it is possible to measure both sub-aortic VTI (gold standard) and sub-pulmonary VTI in one of the two echocardiographic windows described in the literature (parasternal short-axis or subcostal).
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Fluid responsiveness | T0 : baseline T1 : 60 to 90 after passive legs raising manoeuver or mini fluid challenge T2 : within 10 mins after fluid infusion of 500mL of crystalloïds solution
  Echocardiographic measurement of subaortic velocity time integral (AoVTI) in apical 5-chambers view is performed before (T0 = Baseline) and within 10 mins (T2) after fluid administration.
  An increase of 15% or more of AoVTI after fluid administration of 500mL of a crystalloids solution compared to baseline define fluid responsiveness.
Ability of sub-pulmonary VTI variation to predict fluid responsiveness | T0 : Baseline T1 : 60 to 90 after passive legs raising manoeuver or mini fluid challenge T2 : within 10 mins after fluid infusion of 500mL of crystalloïds solution
  The sub-pulmonary VTI variation (in %) between T0 and T1 is mesured with echocardiography from a transthoracic view (short axis parasternal and sub costal views depending of patient's echogenicity)
  Sub-pulmonary VTI variation ability to detect fluid responsiveness is assessed by constructing ROC curves to detect the best cut-off.

SECONDARY OUTCOMES:
Sub-pulmonary VTI values description | T0 : baseline T1 : 60 to 90 after passive legs raising manoeuver or mini fluid challenge T2 : within 10 mins after fluid infusion of 500mL of crystalloïds solution
  To describe values of Sub-pulmonary VTI (cm) during the time frame measured with echocardiography in subcostal view and / or in parasternal short axis view depending of patient's echogenicity.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de réanimation polyvalente - Hopital Nord, Marseille 15
  - Hopital Caremeau Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: Undecided